CLINICAL TRIAL: NCT01066962
Title: An Open-label Randomised Two-year Trial Comparing Two First-line Regimens in HIV-infected Antiretroviral naïve Subjects: Darunavir/r + Tenofovir/Emtricitabine vs. Darunavir/r + Raltegravir (ANRS 143/NEAT 001)
Brief Title: Study of Darunavir/r + Tenofovir/Emtricitabine vs. Darunavir/r + Raltegravir in HIV-infected Antiretroviral naïve Subjects
Acronym: ANRS 143
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: NEAT - European AIDS Treatment Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-015113-44; 2009-015113-44 (EudraCT Number)
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: HIV Infections
Keywords: HIV-infected antiretroviral naïve subjects
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- darunavir/r + tenofovir/emtricitabine (Active Comparator)
  Interventions: Drug: darunavir/r QD + tenofovir/emtricitabine QD (fixed dose combination)
- darunavir/r + raltegravir (Experimental)
  Interventions: Drug: darunavir/ritonavir QD + raltegravir BID

INTERVENTIONS:
Drug: darunavir/ritonavir QD + raltegravir BID — darunavir 800 mg, i.e. 2 tablets of 400 mg once daily (QD)
  ritonavir 100 mg, 1 tablet once daily (QD)
  raltegravir 400 mg, 1 tablet twice daily (BID)
  Arms: darunavir/r + raltegravir
Drug: darunavir/r QD + tenofovir/emtricitabine QD (fixed dose combination) — darunavir 800 mg, i.e. 2 tablets of 400 mg once daily (QD)
  ritonavir 100 mg, 1 tablet once daily (QD)
  tenofovir/emtricitabine 245/200 mg, fixed dose combination, 1 tablet once daily (QD)
  Arms: darunavir/r + tenofovir/emtricitabine

SUMMARY:
The triple therapy darunavir/r + tenofovir/emtricitabine is likely to become a relevant first-line treatment option in the years to come. The dual combination of boosted darunavir + raltegravir is an innovative treatment option that combines two potent new antiretroviral drugs, one of which belongs to a new drug class (integrase inhibitor). The expected efficacy profile of this combination is promising. Moreover, this combination might have a better tolerance profile and has the advantage of sparing the NRTI class.

In the context of tenofovir/emtricitabine currently being a reference backbone in first-line antiretroviral regimens, we hypothesise that, in combination with darunavir/r, raltegravir may be an alternative option if its efficacy is non-inferior to tenofovir/emtricitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed HIV infection
* Age ≥ 18 years
* Written informed consent
* Male patient or non-pregnant, non-lactating female
* No previous treatment with any antiretroviral drugs
* HIV-1 RNA > 1000 copies/ml
* Indication to start an antiretroviral treatment as long as subject has also a CD4 cell count ≤ 500/mm3 either at screening or on a sample taken within 3 months before screening
* No major IAS-USA mutations on genotypic testing at the screening visit or on any historical genotype, if available

Non-inclusion Criteria:

* Woman without effective contraception method (recommended contraception during the trial is mechanical + a second method other than an oral contraceptive)
* Pregnant or breastfeeding woman
* Woman expecting to conceive during the study
* HIV-2 co-infection
* Creatinine clearance < 60 ml/mn (Cockcroft & Gault equation), alkaline phosphatase, ASAT, or ALAT ≥ 5 ULN
* Patient with significant impairment of hepatic function, defined as serum albumin < 2.8 g/dl or INR > 1.7 or presence of ascites, in the absence of another explanation for the abnormal finding
* CD4 > 500/mm3 at screening, except in case of symptomatic HIV disease (defined by conditions qualifying for CDC category B or C) or CD4 ≤ 500/mm3 on a sample taken within 3 months before screening.
* Any major IAS-USA mutation conferring resistance to one or more of reverse transcriptase or protease inhibitors on genotypic testing at screening
* Mycobacteriosis under treatment
* Malignancy requiring chemotherapy or radiotherapy
* Positive HBs Ag
* HCV infection for which specific treatment is ongoing or planned during the first year on trial treatment
* Known hypersensitivity to one of the trial drugs or its excipients
* Contraindicated concomitant treatment
* Anticipated non-compliance with the protocol
* Participation in another clinical trial with an on-going exclusion period at screening
* Subject under legal guardianship or incapacitation
* Subject, who in the opinion of the investigator, is unable to complete the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Time to virologic or clinical failure, as the first occurrence of one of six protocol-defined components | minimum 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François Raffi, Professor, Study Chair — Nantes University Hospital
Locations (77):
- Austria (2):
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Otto Wagner Spital mit Pflegezentrum, Vienna
- Belgium (3):
  - ITZ Antwerpen, Antwerp
  - CHU Saint Pierre, Brussels
  - UZ Gent, Ghent
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Hvidovre Hospital, Hvidovre
- France (18):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Saint André, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Hôpital du Bocage, Dijon
  - Hôpital Pierre Zobda-Quitman, Fort de France
  - CHD de la Roche sur Yon, La Roche-sur-Yon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital de l'Hôtel Dieu, Nantes
  - Hôpital Bichat, Paris
  - Hôpital Européen Georges Pompidou (HEGP), Paris
  - Hôpital La Pitié Salpétrière, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital Foch, Suresnes
  - Hôpital Purpan, Toulouse
  - Hôpital Gustave Dron, Tourcoing
- Germany (8):
  - Gemeinschaftspraxis Jessen-Jessen-Stein, Berlin
  - Med. Universitätsklinik I, Bonn
  - Universitätsklinik Köln, Cologne
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe Universität, Frankfurt
  - Asklepios-Klinik St. Georg, Hamburg
  - ICH study centre, Hamburg
  - Medizinische Hochschule Hannover, Hanover
- Greece (3):
  - Attikon University Hospital, Athens
  - Evaggelismos General Hospital, Athens
  - Laikon General Hospital, Athens
- Saint Laszlo Hospital, Budapest, Hungary
- Ireland (2):
  - Mater Misericordiae, Dublin
  - St James's Hospital, Dublin
- Italy (9):
  - University of Brescia, Brescia
  - Ospedale Santa Maria Annunziata, Florence
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - San Paolo Hospital, Milan
  - Luigi Sacco Hospital, Milan
  - Istituto Naziona e per le Malattie "Lazzaro Spallanzani", Rome
  - Sapienza Universita di Roma, Rome
  - Torvergata University, Rome
  - Ospedale "Amedeo di Savoia", Turin
- Netherlands (3):
  - AMC, Amsterdam
  - Jan van Goyen Medical Center, Amsterdam
  - Rijnstate Hospital, Arnhem
- Hospital of Infectious Diseases of Warsaw, Warsaw, Poland
- Portugal (3):
  - Hospital de Curry Cabral, Lisbon
  - Hospital Santa Maria, Lisbon
  - Hospital de Joaquim Urbano, Porto
- Spain (11):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Clinic, Barcelona
  - Hospital de la Santa Creu I Sant Pau., Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Carlos III, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario La Fe, Valencia
- Sweden (3):
  - Sahlgrenska hospital, Gothenburg
  - Karolinska hospital, Stockholm
  - Venhälsan hospital, Stockholm
- United Kingdom (8):
  - Royal Bournemouth Hospital, Bournemouth
  - Southmead Hospital, Bristol
  - Western General Hospital, Edinburgh
  - Mortimer market centre, London
  - Royal Free Hospital, London
  - Saint Mary's hospital, London
  - Saint Stephen's Centre, London
  - Saint Thomas hospital, London

REFERENCES:
- [Derived] Esteban-Cantos A, Rodriguez-Centeno J, Barruz P, Alejos B, Saiz-Medrano G, Nevado J, Martin A, Gaya F, De Miguel R, Bernardino JI, Montejano R, Mena-Garay B, Cadinanos J, Florence E, Mulcahy F, Banhegyi D, Antinori A, Pozniak A, Wallet C, Raffi F, Rodes B, Arribas JR; NEAT001/ANRS143 Study Group. Epigenetic age acceleration changes 2 years after antiretroviral therapy initiation in adults with HIV: a substudy of the NEAT001/ANRS143 randomised trial. Lancet HIV. 2021 Apr;8(4):e197-e205. doi: 10.1016/S2352-3018(21)00006-0. PMID 33794182
- [Derived] Ammassari A, Stohr W, Antinori A, Molina JM, Schwimmer C, Domingo P, Thalme A, Di Pietro M, Wallet C, Pozniak A, Richert L, Raffi F; NEAT001/ANRS143 Trial Study Group. Patient Self-Reported Adherence to Ritonavir-Boosted Darunavir Combined With Either Raltegravir or Tenofovir Disoproxil Fumarate/Emtricitabine in the NEAT001/ANRS143 Trial. J Acquir Immune Defic Syndr. 2018 Dec 1;79(4):481-490. doi: 10.1097/QAI.0000000000001834. PMID 30365452
- [Derived] Bernardino JI, Mocroft A, Mallon PW, Wallet C, Gerstoft J, Russell C, Reiss P, Katlama C, De Wit S, Richert L, Babiker A, Buno A, Castagna A, Girard PM, Chene G, Raffi F, Arribas JR; NEAT001/ANRS143 Study Group. Bone mineral density and inflammatory and bone biomarkers after darunavir-ritonavir combined with either raltegravir or tenofovir-emtricitabine in antiretroviral-naive adults with HIV-1: a substudy of the NEAT001/ANRS143 randomised trial. Lancet HIV. 2015 Nov;2(11):e464-73. doi: 10.1016/S2352-3018(15)00181-2. Epub 2015 Sep 30. PMID 26520926
- [Derived] Raffi F, Babiker AG, Richert L, Molina JM, George EC, Antinori A, Arribas JR, Grarup J, Hudson F, Schwimmer C, Saillard J, Wallet C, Jansson PO, Allavena C, Van Leeuwen R, Delfraissy JF, Vella S, Chene G, Pozniak A; NEAT001/ANRS143 Study Group. Ritonavir-boosted darunavir combined with raltegravir or tenofovir-emtricitabine in antiretroviral-naive adults infected with HIV-1: 96 week results from the NEAT001/ANRS143 randomised non-inferiority trial. Lancet. 2014 Nov 29;384(9958):1942-51. doi: 10.1016/S0140-6736(14)61170-3. Epub 2014 Aug 4. PMID 25103176